CLINICAL TRIAL: NCT01661959
Title: Scoliosis Outcomes Database Registry
Brief Title: Adolescent Idiopathic Scoliosis Outcomes Database Registry
Acronym: AIS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Setting Scoliosis Straight Foundation (Other)
Collaborators: DePuy Spine (Industry); NuVasive (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007HSGAIS
Record Dates: First submitted 2012-07-10; First posted 2012-08-10 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Multi-center Database Registry; Spinal Deformity; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-Operative
- Operative

SUMMARY:
The purpose of this study is to analyze the long-term outcomes of surgical treatment of idiopathic scoliosis of all curve patterns treated by either anterior or posterior procedures. In addition, to analyze the long-term outcomes of non-operative idiopathic scoliosis.

DETAILED DESCRIPTION:
1. The first aim of this Database Registry is to maintain a prospective multicenter series of patients treated surgically for adolescent idiopathic scoliosis. Patients from multiple scoliosis centers around the U.S., as well as a center in Germany, will be enrolled with comprehensive analysis of the curve pattern being treated, as well as the type of surgery performed. The outcome of each surgical treatment will be analyzed. This will allow the frequency of various curve types to be determined, as well as the frequency of various surgical approaches utilized for each curve pattern.
2. The second aim is to determine if operative outcomes vary based on the surgical approach utilized in scoliosis correction. In this analysis, it is anticipated that specific approaches can be identified to be most appropriate for given scoliotic curve patterns. In addition, the variations within individual curve patterns will be analyzed, as will specific variations in the surgical approach (e.g., distal level of instrumentation, hooks versus screws, hook patterns, etc).
3. The third aim is to develop an algorithm to guide surgical decision making based on a scoliosis curve classification scheme that will allow the surgeon to provide the best overall outcome (radiographic, functional, cosmetic) for a given patient with idiopathic scoliosis.
4. The fourth aim is to evaluate the long-term outcomes of surgical intervention in this patient population.
5. The fifth aim is to maintain a prospective multi-center series of patients with idiopathic scoliosis who have not undergone surgical correction of their deformity. The long-term outcome of this patient population will be compared with the surgical patient population.
6. The sixth aim is to develop a guide to help clinicians make a decision for optimal surgical treatment of AIS curves based on patient-specific 3D information.
7. Factors that may influence intra and post-operative course will also be evaluated. Of particular interest are patient specific factors (curve size, pre op characteristics such as blood work and PFT testing) and their influence on intra-operative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 10 and ≤ 21 years at time of enrollment,
* male or female,
* diagnosis of idiopathic scoliosis for which surgery is recommended to prevent progression of the curvature or to correct trunk disfigurement.
* Curve cobb of any magnitude - operative range
* Spina bifida Oculta is permitted
* Spondylolisthesis and Spondylolysis are permitted, as long as non-operative
* Non-operative idiopathic scoliosis patients:

  * aged ≥ 10 and ≤ 21 years, male or female, curve cobb of ≥ 40º, for whom surgery has been offered and the patient has elected not to proceed with surgery.

OR

- OPTIONAL BY SITE: aged ≥ 10 and ≤ 21 years, male or female, Curve cobb ≥ 30º and skeletally mature (with maturity defined as Age: girls > 14 yrs; Boys > 16 yrs and Risser of ≥ 4 Plus one of the following: Girls 2+ yrs post menarchal, boys shaving regularly, no height change in at least 6 months.

Exclusion Criteria:

* Prior spinal surgery
* MRI abnormalities (including > 4mm of Syrinx and/or Chiari malformation)
* Neuromuscular or other serious co-morbidities
* Thoracogenic or cardiogenic scoliosis
* Associated syndrome or developmental delay
* Unable or unwilling to firmly commit to returning for required follow-up visits

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who present to the investigator's clinic, who meet the inclusion criteria will be offered enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2005-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in radiographic outcome for surgical treatment of idiopathic scoliosis. | 25 years
  Patients are followed up to 25 years post-op.

SECONDARY OUTCOMES:
Change in clinical outcomes for surgical treatment of idiopathic scoliosis. | 25 years
  Patients are followed up to 25 years post-op

CONTACTS AND LOCATIONS:
Overall Officials: Peter O Newton, MD, Principal Investigator — Rady Children's Hospital San Deigo
Locations (14):
- United States (12):
  - Rady Children's Hospital, San Diego, California
  - Nemours Children's Clinic, Wilmington, Delaware
  - Miami Children's Hospital, Miami, Florida
  - John's Hopkins Medical Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington Univ., St. Louis, St Louis, Missouri
  - University Physicians, Camden, New Jersey
  - Scoliosis Associates, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, OH, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
- Canada (2):
  - CHU Saint-Justine Hospital, Montreal
  - British Columbia Children's Hospital, Vancouver

REFERENCES:
- See also: Harms Study Group — http://www.hsg.settingscoliosisstraight.org